CLINICAL TRIAL: NCT00699530
Title: Substrate Metabolism and Insulin Sensitivity in Patients With Hyperprolactinemia Before and After Treatment
Status: Withdrawn | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MM-ISP-20070132
Record Dates: First submitted 2008-05-23; First posted 2008-06-18 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2014-12

CONDITIONS: Hyperprolactinemia; Insulin Resistance
Keywords: Prolactin; Insulin resistance; Glucose tolerance; Body Composition; Substrate metabolism
MeSH Terms: conditions — Hyperprolactinemia; Insulin Resistance | interventions — Cabergoline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, muscle samples, fat samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hyperprolactinemia: Patients recently diagnosed with hyperprolactinemia
  Interventions: Other: Cabergoline

INTERVENTIONS:
Other: Cabergoline — Cabergoline 0,25 - 1,0 mg once a week, controlled by our outpatient clinic. The drug regimen is not influenced by participating in this study.

SUMMARY:
The purpose of this study is to investigate the effects of chronic elevated levels of Prolactin on metabolism and insulin sensitivity by studying patients with hyperprolactinemia before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Age between 18 and 70
* At diagnose a serum prolactin > 200 microgram/l (10 U/l)

Exclusion Criteria:

* Hypothyroidism
* Use of any medication
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recently diagnosed with hyperprolactinemia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Before and after treatment

SECONDARY OUTCOMES:
QoL, body composition, intrahepatic and intramyocellular fat, substrate metabolism, glucose tolerance | Before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L. Jørgensen, Professor MD, Principal Investigator — Aarhus University Hospital, Department of Endocrinology
Locations (1):
- Department of Endocrinology, Aarhus C, Aarhus, Denmark